CLINICAL TRIAL: NCT04432246
Title: Electroencephalography (EEG) Predictors of Repetitive Transcranial Magnetic Stimulation (rTMS) in Obsessive-Compulsive Disorder (OCD): A Preliminary Study
Brief Title: Electroencephalography Predictors of Repetitive Transcranial Magnetic Stimulation in Obsessive-Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, Director, Shanghai Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMHC-OCD-007
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Obsessive Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bilateral SMA (Experimental): Continuous theta burst stimulation (cTBS) stimulation will be applied over the bilateral SMA once a day, 5 days/week, for 4 weeks.
  Interventions: Device: Continuous theta burst stimulation (cTBS)

INTERVENTIONS:
Device: Continuous theta burst stimulation (cTBS) — 50Hz of 90% MT for 3 pulses train over will be repeated at 200ms for the 40s, 600 pulses

SUMMARY:
This study used electroencephalogram (EEG) to predict the efficacy of repetitive transcranial magnetic stimulation (rTMS) in patients with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS), as a relatively mature non-invasive neuromodulation technology, has been recommended for the treatment of patients with refractory OCD in multinational guidelines. However, due to the treatment setting and the patient's feature, nearly half of the patients have no significant changes after rTMS treatment.

In order to better predict the outcome of rTMS and improve the treatment efficiency, this project intends to look for markers that have a predictive effect at baseline or early treatment. Electroencephalogram (EEG) is a cheap and fast method that usually occurs before the symptoms change, thus it is possible to determine whether the patient has responded to the intervention.

In this project, the supplementary motor area (SMA) is selected as the stimulation target. The individual head magnetic resonance image positioning and navigation and rTMS compatible real-time EEG acquisition technology are used to monitor the resting state of EEG and rTMS single pulse stimulation and changes in neural networks before and after treatment. This is a preliminary exploration looking for effective predictive indicators of efficacy in EEG and the relationship between EEG and symptoms changes. In order to lay the foundation for further research and guide clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years old;
* DSM-5 criteria for OCD;
* Y-BOCS total score > or = 16 ->or＝9 yrs education

Exclusion Criteria:

* any additional current psychiatric comorbidity, except for obsessive-compulsive personality disorder serious suicide risk;
* the inability to receive rTMS because of metallic implants, or history of seizures，or history of head injury, or history of neurosurgery;
* any major medical disease;
* pregnancy or nursing of an infant;
* participation in current clinical study;
* current use of any investigational drug;
* TMS/DBS treatment at any point in their lifetime;
* history of long-time use of benzodiazepines

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in symptom improvement assessed by the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Up to 6 months
  It assesses the severity of OCD symptoms. The Y-BOCS scale ranges from 0 to 40, with 0 being no symptoms and 40 being severe.The responder on Y-BOCS is defined as a Y-BOCS decrease at least 35% from the baseline at post-treatment.
EEG biomarkers as predictors of response to rTMS | baseline
  TMS-EEG and resting state EEG will be performed to investigate predictors of response to rTMS in OCD patients. The α, β and δ band power in resting state in each brain area of OCD patients will be recorded and analyzed. Also, in TMS treatment, event related potentials (ERPs) including motor evoked potentials (MEPs) amplitude, I waves, α band power and β band power will be analyzed.

SECONDARY OUTCOMES:
Change in The Beck Depression Inventory (BDI) | Up to 6 months
  It consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression symptoms.
Change in The Beck Anxiety Inventory (BAI) | Up to 6 months
  It is an inventory of anxiety symptoms with 18 items that are rated on a 5-point Likert scale(0 to 4). Total scores range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
Change in The Perceived Stress Scale(PSS) | Up to 6 months
  The Perceived Stress Scale (PSS) has 10 items to assess stress status within four weeks. Items are classified into five levels, from 0 (never) to 4 (very often). Total scores range from 0 to 40. The higher the total score, the stronger the level of stress the patient feels.
Change in Pittsburgh sleep quality index(PSQI) | Up to 6 months
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Change in Obsessive Compulsive Inventory-Revised(OCI-R) | Up to 6 months
  It is an inventory of OCD symptoms with 18 items that are rated on a 5-point Likert scale. Total scores range from 0 to 72, with higher scores indicating more severe OCD symptoms.
Change in Side-effect questionnaire | Up to 6 months
  It consists of 10-item and uses 0 to 3 severity scale to rate the intensity of side effects. Total scores range from 0 to 30, with higher scores indicating more severe side-effect. It also assesses the relation between side-effect and the effects of rTMS using 0 to 4 scale. Total scores range from 0 to 40, with higher score indicating the greater relation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China